CLINICAL TRIAL: NCT02832128
Title: A Pilot Double Blind Placebo Controlled Crossover Study to Explore Possible Benefits of AUT00063, An Oral Modulator of Voltage - Gated Potassium Channels , In Adults Post-lingual Unilateral Cochlear Implant Recipients
Brief Title: Evaluating Possible Improvement in Speech and Hearing Tests After 28 Days of Dosing of the Study Drug AUT00063 Compared to Placebo (QuicKfire)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUT042063; 2015-003929-34 (EudraCT Number)
Record Dates: First submitted 2016-04-04; First posted 2016-07-14 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Hearing Loss; Hearing Impairment
Keywords: Cochlear Implant
MeSH Terms: conditions — Hearing Loss | interventions — AUT00063

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AUT00063 - Placebo (Experimental): AUT00063 (800 mg/day) for 28 days, followed by a 2 to 4 week washout period before commencing the second 28-day dosing period with placebo
  Interventions: Drug: AUT00063; Drug: Placebo
- Placebo - AUT00063 (Experimental): Placebo for 28 days, followed by a 2 to 4 week washout period before commencing the second 28-day dosing period with AUT00063 (800 mg/day)
  Interventions: Drug: AUT00063; Drug: Placebo

INTERVENTIONS:
Drug: AUT00063 — 4 capsules of 200 mg AUT00063, to take orally with food for 4 weeks
Drug: Placebo — 4 capsules of placebo, to take orally with food for 4 weeks

SUMMARY:
The objective of this pilot study is to explore whether repeat doses of AUT00063 can provide an indication of improvement in performance of tests across a battery of speech and hearing assessments in cochlear implant users.

DETAILED DESCRIPTION:
Reduced activity at certain sites in the brain called "voltage-gated potassium channels", has been linked to hearing problems. The study drug, AUT00063, has been developed to help improve the recognition of speech by aiming to improve the action of the voltage-gated potassium channels in the hearing pathways in the brain and so help to treat the hearing problem.

The main purpose of this study is to find out whether AUT00063 can improve the understanding of speech after 28 days of treatment compared with a placebo (dummy drug which does not contain the study drug) in patients who have received a cochlear implant (CI) for post-lingual deafness.

Efficacy will be investigated through a number of assessments including speech recognition testing, parameters of central auditory processing measured using tests that involve direct stimulation via the CI, and questionnaires.

Safety assessments will also be conducted throughout the study including physical examinations, ECGs and blood sampling.

It is planned that up to 20 people who have received a cochlear implant within the last 9 to 36 months will take part in the study. The people will be recruited from around 4 hospital sites in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years.
* Native English speaking.
* Received a unilateral cochlear implant within the last 9 to 48 months for post-lingual deafness.
* Less than optimal speech perception at the time of enrolment (defined as a score of 25% to 95% for Bamford-Kowal-Bench (BKB) sentences.
* Fully trained and optimised at the time of enrolment.
* CI device working satisfactorily and no interventions in the 4 weeks prior to the first dose of study medication.
* Signed and dated informed consent.

Exclusion Criteria:

* Not able to understand and comply with the requirements of the study.
* CI undertaken primarily for the management of severe tinnitus.
* Moderate or severe depression or generalised anxiety.
* Currently taking or planning to take medications that are prohibited by the study protocol.
* History of important cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases deemed clinically significant.
* Clinically significant ECG abnormality or prolonged QT interval.
* Screening laboratory safety test results outside the normal ranges that are deemed to be clinically significant by the investigator.
* Any acute disabling illness.
* Clinically significant alcohol or drug abuse.
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives of the investigational drug.
* For women: Pregnant or nursing.
* For men and women: Not willing or able to use adequate methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Speech recognition tests | 10 - 12 weeks
  To compare % scores on a battery of speech tests after 28 days of AUT00063 compared to baseline and placebo

SECONDARY OUTCOMES:
Direct stimulation tests | 10 - 12 weeks
  To compare rate discrimination and gap detection thresholds after 28 days of AUT00063 compared to baseline and placebo
To further investigate the safety and tolerability profile of repeat administration of AUT00063 | up to 15 weeks
  To investigate the safety and tolerability of AUT00063 by assessing vital signs, physical examination, laboratory exams and ECG

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel R Saeed, MD, FRCS (ORL), Principal Investigator — Royal National Throat, Nose and Ear Hospital
Locations (4):
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal National Throat, Nose and Ear Hospital, London
  - Manchester Royal Infirmary, Manchester